CLINICAL TRIAL: NCT01212536
Title: Randomised Controlled Trial of the Airtraq Optical Laryngoscope and Conventional Laryngoscopy in Children
Brief Title: Airtraq Versus Conventional Laryngoscopy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Michelle White, Consultant in Paediatric Anaesthesia and Critical Care, University Hospitals Bristol and Weston NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CH/2009/3387
Record Dates: First submitted 2010-07-15; First posted 2010-09-30 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Children; General Anesthesia; Intubation
Keywords: children; intubation; laryngoscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional (No Intervention): conventional laryngoscopy for intubation
- Airtraq (Experimental): laryngoscopy with Airtraq for intubation
  Interventions: Device: Airtraq laryngoscopy

INTERVENTIONS:
Device: Airtraq laryngoscopy — laryngoscopy and intubation
  Arms: Airtraq

SUMMARY:
The investigators aim to compare the new paediatric Airtraq indirect optical laryngoscope with conventional direct laryngoscopy for tracheal intubation in a randomised crossover study during routine anaesthesia. The investigators hypothesise that the Airtraq is as good as conventional laryngoscopy for tracheal intubation of infants and children. This will be an equivalence rather than a non-inferiority study.

ELIGIBILITY:
Inclusion Criteria:

* All children less than 6 years of age, in whom a size 2.5 - 5.5 tracheal tube would be considered suitable.
* Classified by the American Society of Anesthesiology (ASA) as grade 1-3.
* Scheduled for surgery under general anaesthesia, and in whom tracheal intubation and neuromuscular blocking drugs are planned to be used.

Exclusion Criteria:

* inability of patient or parents to understand the study or consent process
* known or suspected difficult airway
* ASA 4 and above

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
time taken to successful intubation | 30 mins
  The primary outcome measure will be time taken to successful intubation. This will be recorded by a second operator using a handheld stopwatch or wall clock with second hand. Time will commence when the intubation device is handed to the anaesthetist, and stopped after the first successful inflation of the lungs (first upstroke of capnography trace).

SECONDARY OUTCOMES:
Grade of laryngoscopy | 30 mins
POGO score | 30 mins
VAS ease of intubation | 30 mins
evidence of traumatic intubation | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol Childrens hospital, Bristol, Bristol, United Kingdom